CLINICAL TRIAL: NCT03290937
Title: Phase I Clinical Trial Evaluating the Safety and Response With PF-05082566, Cetuximab, and Irinotecan in Patients With Advanced Colorectal Cancer
Brief Title: Utomilumab, Cetuximab, and Irinotecan Hydrochloride in Treating Patients With Metastatic Colorectal Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017-0180; NCI-2018-01036 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2017-0180 (Other: M D Anderson Cancer Center); P30CA016672 (NIH)
Record Dates: First submitted 2017-09-20; First posted 2017-09-25 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Metastatic Colorectal Carcinoma; Stage IV Colorectal Cancer AJCC v8; Stage IVA Colorectal Cancer AJCC v8; Stage IVB Colorectal Cancer AJCC v8; Stage IVC Colorectal Cancer AJCC v8
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Cetuximab; Irinotecan; utomilumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (irinotecan hydrochloride, cetuximab, utomilumab) (Experimental): Patients receive irinotecan hydrochloride IV over 90 minutes and cetuximab IV over 1-2 hours on days 1 and 15, and utomilumab IV over 1 hour on day 2. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Cetuximab; Drug: Irinotecan Hydrochloride; Other: Pharmacodynamic Study; Biological: Utomilumab

INTERVENTIONS:
Biological: Cetuximab — Given IV
  Other Names: Cetuximab Biosimilar CDP-1; Cetuximab Biosimilar CMAB009; Cetuximab Biosimilar KL 140; Chimeric Anti-EGFR Monoclonal Antibody; Chimeric MoAb C225; Chimeric Monoclonal Antibody C225; Erbitux; IMC-C225
Drug: Irinotecan Hydrochloride — Given IV
  Other Names: Campto; Camptosar; Camptothecin 11; Camptothecin-11; CPT 11; CPT-11; Irinomedac; Irinotecan Hydrochloride Trihydrate; Irinotecan Monohydrochloride Trihydrate; U-101440E
Other: Pharmacodynamic Study — Correlative studies
  Other Names: PHARMACODYNAMIC
Biological: Utomilumab — Given IV
  Other Names: PF 05082566; PF 5082566; PF-05082566; PF-2566

SUMMARY:
This phase I trial studies the best dose and side effects of irinotecan hydrochloride when given with utomilumab and cetuximab in treating patients with colorectal cancer that has spread to other places in the body (metastatic). Monoclonal antibodies, such as utomilumab and cetuximab, may interfere with the ability of tumor cells to grow and spread. Drugs used in chemotherapy, such as irinotecan hydrochloride, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving utomilumab, cetuximab, and irinotecan hydrochloride may work better in treating patients with colorectal cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate maximal tolerated dose (MTD), and recommended phase 2 dose (RP2D) of the combination of utomilumab (PF-05082566), cetuximab and irinotecan hydrochloride (irinotecan) (PCI) in patients with metastatic colorectal cancer refractory to standard therapy. (Dose escalation) II. To determine the antitumor activity overall response rate (ORR) by immune-related Response Evaluation Criteria in Solid Tumors (irRECIST) of the study regimen specifically in patients with advanced colorectal cancer who are RAS-RAF wild type (WT) (Arm A) or RAS mutant (Arm B). (Dose expansion)

SECONDARY OBJECTIVES:

I. To evaluate overall safety profile. II. To evaluate the anti-tumor activity. III. To evaluate pharmacodynamics (PD) biomarkers expressed by peripheral blood mononuclear cells (PBMC) and tissue samples.

IV. To characterize serum biomarkers linked to immunomodulation and cytokine release.

V. To assess markers of T and natural killer (NK) cell phenotype (such as CD3, CD4, CD8, FoxP3, CD14, CD33, CCR7, CD45RO, CD16, CD56, CD69, CD25, or VCAM1), TNF alpha, IFN gamma, IL10, IL-8, IL-6, IL-4, IL-2, IL-1b, or IL-12p70, CD127, Ki67, eomesodermin, KLRG1, CD14, CD33, human leukocyte antigen- D related (HLA-DR), CD16, CD56, granzyme B, CD68, PD-1, CD11c, sCD137, and 4-1BB.

OUTLINE: This is a dose escalation study of irinotecan hydrochloride.

Patients receive irinotecan hydrochloride intravenously (IV) over 90 minutes and cetuximab IV over 1-2 hours on days 1 and 15, and utomilumab IV over 1 hour on day 2. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically and or cytologically confirmed metastatic colorectal cancer
* Patients must have a wild type or mutated RAS tumor status known prior to enrollment
* Metastatic colorectal cancer patients have progressed following at least one line of fluorouracil (5-FU)-based chemotherapy
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2
* Patients must have measurable disease per irRECIST criteria for part 2 (dose expansion)
* Absolute neutrophil count (ANC) >= 1.0 x 10^9/L (1,000/uL)
* Platelet count >= 75 x 10^9/L (75000/L)
* Hemoglobin >= 8.0 g/dL (>= 5.0 mmol/L)
* Patients must be transfusion independent (i.e., no blood product transfusions for a period of at least 14 days prior to screening)
* Serum creatinine < 2 x upper limit of normal (ULN) or estimated creatinine clearance > 30 ml/min as calculated using the method standard for the institution
* Total serum bilirubin < 1.5 x ULN, unless the patient has documented Gilbert syndrome
* Aspartate and Alanine Aminotransferase (AST and ALT) < 3 x ULN
* Left ventricular ejection fraction (LVEF) that is greater than 40%, or the absence of New York Heart Association (NYHA) classification of greater than stage II congestive heart failure
* Resolved acute effects of any prior therapy to baseline severity or grade =< 2 Common Terminology Criteria for Adverse Events (CTCAE) version (v.) 4.03 except for adverse events (AEs) not constituting a safety risk by investigator judgment
* Serum or urine pregnancy test (for females of childbearing potential) negative at screening and at the baseline visit (before the patient may receive the investigational product)
* Male and female patients of childbearing potential and at risk for pregnancy must agree to use two highly effective methods of contraception throughout the study and for at least 90 days after the last dose of assigned treatment. Female patients who are not of childbearing potential (permanently sterilized or postmenopausal; i.e., meet at least one of the following criteria):

  * Have undergone a documented hysterectomy and/or bilateral oophorectomy; or
  * Have medically confirmed ovarian failure; or
  * Achieved postmenopausal status, defined as follows: cessation of regular menses for at least 12 consecutive months with no alternative pathological or physiological cause; status may be confirmed by having a serum follicle stimulating hormone (FSH) level within the laboratory's reference range for postmenopausal women
* High microsatellite instability (MSI-H) colorectal cancer patients must have received an approved PD-1 targeted agent prior to enrolling in this trial
* Evidence of a personally signed and dated informed consent document indicating that the patient has been informed of all pertinent aspects of the study
* Co-consent for protocol LAB10-0982
* Willingness and ability to comply with the study scheduled visits, treatment plans, laboratory tests and other procedures

Exclusion Criteria:

* Patients with known symptomatic brain metastases requiring steroids. Patients with previously diagnosed brain metastases are eligible if they are asymptomatic or have completed their treatment and have recovered from the acute effects of radiation therapy or surgery prior to the start of study medication, have discontinued corticosteroid treatment for these metastases for at least 4 weeks and are neurologically stable
* Patient has had any treatment specific for tumor control within 3 weeks of dosing, or for investigational drugs and cytotoxic agents, within 5 half-lives or 3 weeks, whichever is shorter
* Patients receiving any medications or substances that are strong inhibitors or inducers of CYP3A4 complex. Lists including medications and substances known or with the potential to interact with the CYP3A4 isoenzymes
* Prior therapy with a compound of the same mechanism as PF-05082566 (immunomodulation of 4-1BB)
* Major surgery within 28 days of starting study treatment
* Radiation therapy within 14 days of starting study treatment
* Autoimmune disorders (e.g., Crohn's disease, rheumatoid arthritis, scleroderma, systemic lupus erythematosus) and other diseases that compromise or impair the immune system except patients who have grade 1 psoriasis (in remission or controlled with topical steroids) or mild degree of autoimmune thyroiditis that are controlled with medications
* Active and clinically significant bacterial, fungal or viral infection including hepatitis B (HBV), hepatitis C (HCV), known human immunodeficiency virus (HIV) or acquired immunodeficiency syndrome (AIDS)-related illness (HIV testing is not required)
* Unstable or serious concurrent medical conditions in the previous 6 months, e.g., pancreatitis, severe/unstable angina, prolonged QT interval corrected by Fridericia's formula (QTcF) > 470 msec (calculated as average of triplicate readings, taken no greater than 2 minutes apart, and no history of torsades de pointes or symptomatic corrected QT [QTc] abnormality), symptomatic congestive heart failure, myocardial infarction and/or pulmonary hypertension, ongoing maintenance therapy for life-threatening ventricular arrhythmia, stroke, and uncontrolled major seizure disorder
* Concurrent active malignancy other than non-melanoma skin cancer or carcinoma in situ of the cervix
* Patients who are pregnant or breastfeeding
* Patients with intolerance to or who have had a severe allergic or anaphylactic reaction to antibodies or infused therapeutic proteins, or patients who have had a severe allergic or anaphylactic reaction to any of the substances included in the study drug (including excipients)
* Other severe acute or chronic medical or psychiatric condition, including recent (within the past year) or active suicidal ideation or behavior, or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the patient inappropriate for entry into this study

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2017-12-27 (Actual); Primary Completion 2025-12-30 (Actual); Study Completion 2025-12-30 (Actual)

PRIMARY OUTCOMES:
Recommended phase 2 dose of irinotecan hydrochloride (Dose escalation) | Up to 4 years
  A modified 3+3 design will be used to determine the maximum tolerated dose.
Objective response rate (Dose expansion) | Up to 4 years
  Assessed by using the immune-related Response Evaluation Criteria in Solid Tumors (irRECIST).

SECONDARY OUTCOMES:
Incidence of adverse events | Up to 4 years
  Characterized by type, frequency, severity (as graded by National Cancer Institute [NCI] Common Terminology Criteria for Adverse Events [CTCAE] version [v.]4.03), timing, seriousness and relationship to study therapy utolimumab (PF-05082566); Laboratory abnormalities as characterized by type, frequency, severity (as graded by NCI CTCAE v.4.03) and timing.
Progression free survival | Up to 4 years
  Will be analyzed using Kaplan-Meier methods and descriptive statistics.
Overall survival | Up to 4 years.
  Will be analyzed using Kaplan-Meier methods and descriptive statistics.
Overall response rate | Up to 4 years
Duration of response | Up to 4 year

CONTACTS AND LOCATIONS:
Overall Officials: David S Hong, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

DOCUMENTS (1):
  • Informed Consent Form (2020-05-18): https://cdn.clinicaltrials.gov/large-docs/37/NCT03290937/ICF_000.pdf